CLINICAL TRIAL: NCT02975505
Title: Pilot to Examine Risk and Feasibility of Remote Management of BP From CKD Through ESRD
Acronym: PERFORMANCE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to challenges in recruitment and visits during COVID
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-20978
Record Dates: First submitted 2016-11-22; First posted 2016-11-29 (Estimated); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Chronic Kidney Disease; Bloodpressure; Hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strict SBP Target (Experimental): Target Systolic Home Blood Pressure <120 mm Hg
  Interventions: Other: Strict blood pressure control
- Usual SBP Target (No Intervention): Target Systolic Home Blood Pressure 130-140 mm Hg

INTERVENTIONS:
Other: Strict blood pressure control — Systolic Blood Pressure Target < 120 mm Hg (measured at home)
  Arms: Strict SBP Target

SUMMARY:
The transition from chronic kidney disease (CKD) to end-stage renal disease ESRD is a vulnerable and challenging period of time for patients and providers. Suboptimal control of blood pressure is known to be common in patients with the advanced stages of CKD, and may contribute to their elevated risk of progression to ESRD, cardiovascular morbidity, and mortality. This proposal is a pilot randomized controlled trial designed to test whether intensive home blood pressure lowering is feasible and safe in patients with advanced CKD as they transition to ESRD.

DETAILED DESCRIPTION:
The transition from advanced chronic kidney disease (CKD), when estimated glomerular filtration rate (eGFR) is <=30 mL/min/1.73m2, to end-stage renal disease (ESRD) represents a vulnerable period, when multiple physiologic and psychosocial changes occur as patients prepare for either dialysis or kidney transplant. This study is a pilot randomized controlled trial to test the safety and feasibility of studying strict versus usual BP control in a population of patients with advanced CKD (eGFR <=30 mL/min/1.73m2), including those with diabetes. For this pilot study, we will randomize 120 patients with advanced CKD who have elevated BP to either a home SBP target of <120 mm Hg (intervention group) versus usual care (130-140 mmHg).

ELIGIBILITY:
Inclusion Criteria:

Adults ≥16 years of age who meet the eGFR eligibility criteria, which will be determined based on whether participants have

1. at least two eGFR in the last three months that are <=30 mL/min/1.73m2 or
2. prior diagnosis of CKD (per electronic chart review) and at least one eGFR <=30 mL/min/1.73m2
3. history of hypertension
4. mid-arm circumference between 22-37cm (BP cuff size limitation) and be able to provide consent to participate in our study.

Exclusion criteria

Those who:

* are or are planning to become pregnant, due to inability to take multiple classes of anti-hypertensive agents
* are marginally housed, due to concerns regarding routine follow-up
* are actively participating in a different interventional trial that may affect blood pressure
* are unwilling to consent to participate
* institutionalized individuals or prisoners
* are actively abusing illicit drugs or alcohol
* have a history of poor or doubtful compliance (e.g., frequently missed appointments)
* have office SBP >170 mmHg
* are already taking >5 anti-hypertensive medications (any classes, including diuretics) have cognitive impairment prohibiting participation in the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2021-07-18 (Actual); Study Completion 2021-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Hsu, MD MAS, Principal Investigator — University of California, San Francisco; Elaine Ku, MD MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ku E, Copeland TP, McCulloch CE, Seth D, Carlos CA, Cho K, Malkina A, Lo LJ, Hsu RK. Intensive Home Blood Pressure Lowering in Patients With Advanced CKD. Am J Kidney Dis. 2025 Mar;85(3):320-328. doi: 10.1053/j.ajkd.2024.08.010. Epub 2024 Oct 18. PMID 39427725

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual SBP Target | Strict SBP Target
Started | 42 | 66
Month 4 | 38 | 61
Completed (Month 8) | 34 | 59
Not Completed | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual SBP Target | Strict SBP Target | Total
Number analyzed (Participants) | 42 | 66 | 108
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [43 to 70] | 53 [33 to 62] | 56 [38 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 29 | 47
  Male | 24 | 37 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 12 | 15
  Not Hispanic or Latino | 39 | 54 | 93
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian or Pacific Islander | 14 | 21 | 35
  Black | 3 | 6 | 9
  Native American | 1 | 1 | 2
  Other | 3 | 12 | 15
  White | 21 | 26 | 47
Clinic systolic blood pressure [Median (Inter-Quartile Range); unit: mmHg] | 135 [125 to 151] | 135 [120 to 150] | 135 [124 to 151]
Clinic diastolic blood pressure [Median (Inter-Quartile Range); unit: mmHg] | 79 [72 to 85] | 81 [72 to 87] | 79 [72 to 86]
Diabetes [Count of Participants; unit: Participants] | 14 | 19 | 33
Baseline eGFR [Median (Inter-Quartile Range); unit: mL/min/1.73 m2] | 24 [17 to 27] | 24 [19 to 27] | 24 [18 to 27]
Urine protein/creatinine ratio [Median (Inter-Quartile Range); unit: g/g] | 1 [1 to 3] | 1 [1 to 3] | 1 [1 to 3]
History of heart failure [Count of Participants; unit: Participants] | 3 | 4 | 7
History of acute coronary syndrome [Count of Participants; unit: Participants] | 2 | 5 | 7
History of Smoking [Count of Participants; unit: Participants]
  Never | 23 | 37 | 60
  Former | 18 | 27 | 45
  Current | 1 | 2 | 3
Insurance [Count of Participants; unit: Participants]
  Medicare | 20 | 25 | 45
  Medicaid | 3 | 9 | 12
  Private | 19 | 32 | 51

OUTCOME MEASURES:

1. Primary Outcome: Achieved Clinic Systolic Blood Pressure
Description: Achieved clinic SBP at month 12
Time Frame: At month 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Usual SBP Target | Strict SBP Target
Number analyzed (Participants) | 42 | 66
mmHg | 138.2 (5.3) | 124.7 (3.8)

2. Primary Outcome: Difference in Clinic SBP Between the Two Arms
Description: Incorporating achieved mean SBP data between months 4-12
Time Frame: Months 4-12
Population: Difference is measured between months 4-12
Measure: Mean (95% Confidence Interval); unit: mmHg
Groups:
- Overall Trial: Mean difference (less intensive - intensive)
Arm/Group | Overall Trial
Number analyzed (Participants) | 108
mmHg | 11.7 [7.5 to 16]
Statistical Analysis 1: Comparison: Overall Trial; Test type: Superiority; p < 0.05, Mixed Models Analysis; beta = 11.7, 95% CI 2-sided [7.5 to 16]

3. Primary Outcome: Hyperkalemia, Syncope, Falls, ESKD
Description: Potassium >=6 or self-reported syncope or falls or discharge diagnosis of acute kidney injury from emergency room or hospitalization
Time Frame: Months 0-12
Measure: Count of Participants; unit: Participants
Groups:
- Strict SBP Control: Target Systolic Home Blood Pressure <120 mm Hg
  Strict blood pressure control: Systolic Blood Pressure Target < 120 mm Hg (measured at home)
- Usual SBP Control: Target Systolic Home Blood Pressure 130-140 mm Hg
Arm/Group | Strict SBP Control | Usual SBP Control
Number analyzed (Participants) | 66 | 42
Participants
  Hyperkalemia | 2 | 2
  Syncope | 1 | 3
  Falls | 9 | 7
  Dialysis or (re)-transplant | 3 | 0

4. Secondary Outcome: Screening to Enrollment Ratio
Description: This is the number of potential participants screened as eligible to the number who agree to enroll
Time Frame: From baseline entry through the end of Year 3 of study
Population: Number of participants screened to enroll 1 participant
Measure: Number; unit: participants
Groups:
- Overall Trial: Screening to enrollment ratio
Arm/Group | Overall Trial
Number analyzed (Participants) | 724
participants | 108

5. Other Pre Specified Outcome: Difference in Achieved SBP
Description: Clinic
Time Frame: Between month 4 after baseline and year 4 of study
Measure: Mean (95% Confidence Interval); unit: mmHg
Groups:
- Difference in Clinic SBP: Between month 4 and study end
Arm/Group | Difference in Clinic SBP
Number analyzed (Participants) | 108
mmHg | 12.5 [9 to 16.1]
Statistical Analysis 1: Comparison: Difference in Clinic SBP; Test type: Superiority; p = 0.05, Mixed Models Analysis; beta = 12.5, 95% CI 2-sided [8 to 16]

6. Other Pre Specified Outcome: Hyperkalemia, Syncope, Falls, ESKD
Description: Potassium >=6 or self-reported syncope or falls or discharge diagnosis or need of dialysis or retransplantation
Time Frame: Between month 4 after baseline and year 4 of study
Measure: Count of Participants; unit: Participants
Arm/Group | Strict SBP Control | Usual SBP Control
Number analyzed (Participants) | 66 | 42
Participants
  Hyperkalemia | 2 | 2
  Syncope | 1 | 4
  Falls | 11 | 8
  Dialysis or (re)-transplant | 14 | 4

ADVERSE EVENTS:
Time Frame: Between baseline and year 4 of study
Description: The study team collected adverse event information from the participants weekly.
Arm/Group | Strict SBP Target | Usual SBP Target
All-Cause Mortality (participants affected / at risk) | 5/66 | 2/42
Serious Adverse Events (participants affected / at risk) | 30/66 | 22/42
Other Adverse Events (participants affected / at risk) | 18/66 | 10/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Strict SBP Target (N=66) | Usual SBP Target (N=42)
All-cause hospitalization (Investigations) | 30 | 22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Strict SBP Target (N=66) | Usual SBP Target (N=42)
Acute kidney injury or ER visit (Renal and urinary disorders) | 18 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2025-02-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT02975505/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT02975505/SAP_001.pdf